CLINICAL TRIAL: NCT01932320
Title: An Open Label Study to Investigate the Relative Bioavailability, Food Effect and Effect of Ketoconazole on the Rate and Extent of Absorption of Solid Dosage Formulation(s) of JNJ-40411813
Brief Title: A Study to Evaluate the Relative Bioavailability, Food Effect and Effect of Ketoconazole on the Rate and Extent of Absorption of Solid Dosage Formulation(s) of JNJ-40411813
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016765; 40411813EDI1004 (Other: Johnson & Johnson Pharmaceutical Research & Development); 2009-016638-28 (EudraCT Number)
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Healthy; Relative Bioavailability; Food effect; JNJ-40411813; Positive allosteric modulator; Solid Dosage Formulation of JNJ-40411813; Ketoconazole
MeSH Terms: interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): Participants will receive single dose of all the 3 formulations of JNJ-40411813 (Formulation A: hard gelatin capsule filled with beads; Formulation B: immediate release tablet, and Formulation C: Nanosuspension formulation) without food in 3 periods (Period 1, Period 2, and Period 3). The sequences will be based on a computer-generated randomization schedule prepared by the sponsor before the study. Each period will be separated by a wash out period (no treatment) of at least 1 week.
  Interventions: Drug: JNJ-40411813: Formulation A; Drug: JNJ-40411813: Formulation B; Drug: JNJ-40411813: Formulation C
- Part 2 (Experimental): Participants will receive single dose of the selected solid dose formulation of JNJ-40411813 (Formulation A or Formulation B) from Part 1 without food and with food in 2 periods (Period 1 and Period 2). The sequences will be based on a computer generated randomization schedule prepared by the sponsor before the study. Each period will be separated by a wash out period of at least 1 week.
  Interventions: Drug: JNJ-40411813: Formulation A; Drug: JNJ-40411813: Formulation B
- Part 3 (Experimental): Participants will receive single dose of the selected solid dose formulation of JNJ-40411813 (Formulation A or Formulation B) from Part 1 on two occasions (Day 1 and Day 10) without food along with ketoconazole from Day 6 to Day 14 with food.
  Interventions: Drug: JNJ-40411813: Formulation A; Drug: JNJ-40411813: Formulation B; Drug: Ketoconazole

INTERVENTIONS:
Drug: JNJ-40411813: Formulation A — Participants will receive JNJ-40411813 100 mg hard gelatin capsule orally (by mouth) as a single dose for Part 1 (Period 1, Period 2, and Period 3). If selected this formulation from Part 1, participants will receive this formulation at the dose of 50 mg to 150 mg orally without food and with food in Part 2 (Period 1, Period 2); and at the dose of 50 mg to 150 mg orally without food on Day 1 and Day 10 in Part 3.
Drug: JNJ-40411813: Formulation B — Participants will receive JNJ-40411813 100 mg immediate release tablet orally as a single dose for Part 1 (Period 1, Period 2, and Period 3). If selected this formulation from Part 1, participants will receive this formulation at the dose of 50 mg to 150 mg orally without food and with food in Part 2 (Period 1, Period 2); and at the dose of 50 mg to 150 mg orally without food on Day 1 and Day 10 in Part 3.
Drug: JNJ-40411813: Formulation C — Participants will receive JNJ-40411813 100 mg nanosuspension orally as a single dose for Part 1 (Period 1, Period 2, and Period 3).
  Arms: Part 1
Drug: Ketoconazole — Participants will receive ketoconazole 200 mg tablet orally twice daily with food from Day 6 to Day 14 in Part 3.
  Arms: Part 3

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of a single dose of two solid dose formulations relative to a nanosuspension formulation of JNJ-40411813 (Part 1); to evaluate the effect of a high-fat/high-calorie breakfast on the rate and extent of absorption of the selected JNJ-40411813 solid dose formulation from Part 1 (Part 2); and to explore the influence of a potent inhibitor of CYP3A4, ketoconazole, on the rate and extent of absorption of the selected JNJ-40411813 solid dose formulation from Part 1 (Part 3).

DETAILED DESCRIPTION:
This is an open-label (both physician and participants know the identity of the intervention) and single centre study. This study will be conducted in 3 parts (Part 1, Part 2, and Part 3). The study consists of 3 phases including, the screening phase (within 21 days prior to the start of study medication), treatment phase (Part 1: 20 days; Part 2: 12 days; Part 3: 16 days), and the follow-up phase (Part 1 and Part 2: approximately 14 days after the last administration of study medication and Part 3: 14 days after the last administration of ketaconazole). Approximately 36 participants will be enrolled in the study (12 participants in each part). Part 1 is randomized (study medication is assigned by chance) and 3-way cross-over (method used to switch participants from one treatment arm to another in a clinical study) part of the study. Participants in Part 1 will be randomly assigned to 1 of 3 treatment sequences (Period 1, Period 2, and Period 3) to receive single dose of 3 formulations of JNJ-40411813 (Formulation A: hard gelatin capsule filled with beads; Formulation B: immediate release tablet; and Formulation C: nanosuspension formulation) without food. Each period will be separated by a wash out period (no treatment) of at least 1 week. Part 2 is randomized and 2-way cross-over part of the study. Participants in Part 2 will be randomly assigned 1 of 2 treatment sequences (Period 1 and Period 2) to receive single dose of the selected solid dose formulation of JNJ-40411813 from Part 1 without food and with food separated by a wash out period of at least 1 week. Part 3 is single-arm sequential (carried out in a staged approach) part of the study. Participants in Part 3 will receive single dose of the selected solid dose formulation of JNJ-40411813 from Part 1 on two occasions (Day 1 and Day 10) without food along with ketoconazole from Day 6 to Day 14 with food. Safety will be evaluated by the assessment of adverse events, vital signs, physical examination, 12-lead electrocardiogram, and clinical laboratory tests which will be monitored throughout the study. The total duration of study participation for a participant will be 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index (BMI) between 18 and 30 kg/m2 (BMI is calculated as weight [kilogram] divided by square of height [meter])
* Non-smoker (not smoked for 3 months prior to screening)

Exclusion Criteria:

* Clinically significant abnormal values for laboratory tests and abnormal physical examination
* History of or current significant unstable medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection
* History of epilepsy or fits or unexplained black-outs and significant history of or current psychiatric or neurological illness
* Serology positive for hepatitis B surface antigen, hepatitis C antibodies or HIV antibodies at screening
* Positive urine screen for drugs of abuse and positive alcohol breath test at screening or start of study medication
* Clinically significant acute illness within 7 days prior to start of study medication
* Use of any prescription medication or over-the-counter medication (not including paracetamol), or herbal medication within 2 weeks of start of study medication

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration of JNJ-40411813 | 1 hour predose to 96 hours postdose (for Part 1 and Part 2 [after each single-dose administration]) and 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for 3 formulations of JNJ-40411813: Formulation A: hard gelatin capsule filled with beads; Formulation B: immediate release tablet; and Formulation C: nanosuspension formulation.
Time to reach the peak plasma concentration of JNJ-40411813 | 1 hour predose to 96 hours postdose (for Part 1 and Part 2 [after each single-dose administration]) and 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for 3 formulations of JNJ-40411813: Formulation A: hard gelatin capsule filled with beads; Formulation B: immediate release tablet; and Formulation C: nanosuspension formulation.
Area under the plasma concentration of JNJ-40411813-time curve from 0 to t hours post dosing | 1 hour predose to 96 hours postdose (for Part 1 and Part 2 [after each single-dose administration]) and 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for 3 formulations of JNJ-40411813: Formulation A: hard gelatin capsule filled with beads; Formulation B: immediate release tablet; and Formulation C: nanosuspension formulation.
Area under the plasma concentration of JNJ-40411813 time curve from 0 to infinity post dosing | 1 hour predose to 96 hours postdose (for Part 1 and Part 2 [after each single-dose administration]) and 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for 3 formulations of JNJ-40411813: Formulation A: hard gelatin capsule filled with beads; Formulation B: immediate release tablet; and Formulation C: nanosuspension formulation.
Elimination rate constant of JNJ-40411813 | 1 hour predose to 96 hours postdose (for Part 1 and Part 2 [after each single-dose administration]) and 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for 3 formulations of JNJ-40411813: Formulation A: hard gelatin capsule filled with beads; Formulation B: immediate release tablet; and Formulation C: nanosuspension formulation.
Terminal half-life of JNJ-40411813 | 1 hour predose to 96 hours postdose (for Part 1 and Part 2 [after each single-dose administration]) and 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for 3 formulations of JNJ-40411813: Formulation A: hard gelatin capsule filled with beads; Formulation B: immediate release tablet; and Formulation C: nanosuspension formulation.
Relative bioavailability of JNJ-40411813 | 1 hour predose to 96 hours postdose (for Part 1 and Part 2 [after each single-dose administration]) and 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for 3 formulations of JNJ-40411813: Formulation A: hard gelatin capsule filled with beads; Formulation B: immediate release tablet; and Formulation C: nanosuspension formulation.
Cumulative amount of JNJ-40411813 excreted in urine | 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for solid formulation of JNJ-40411813.
Renal clearance of JNJ-40411813 | 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for solid formulation of JNJ-40411813.
Fraction of JNJ-40411813 excreted in urine until time 't' | 1 hour predose to 120 hours postdose (for Part 3 [after each single-dose administration])
  This pharmacokinetics parameter will be analyzed for solid formulation of JNJ-40411813.

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 8 weeks (for Part 1, Part 2, and Part 3)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Antwerp, Belgium